CLINICAL TRIAL: NCT04664036
Title: Prevalence, Incidence and Characteristics of NAFLD/NASH in Type 1 Diabetes Mellitus Obtained Via a Non-invasive Screening Protocol
Brief Title: Prevalence, Incidence and Characteristics of NAFLD/NASH in Type 1 Diabetes Mellitus
Acronym: NAFLDIA1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Christophe De Block, Prof. dr. Christophe De Block, University Hospital, Antwerp
Other Study IDs: 18/32/361
Record Dates: First submitted 2020-11-04; First posted 2020-12-11 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: NAFLD; Type 1 Diabetes; Cardiovascular Diseases
Keywords: NAFLD; type 1 diabetes; cardiovascular disease; insulin resistance
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 1; Cardiovascular Diseases; Insulin Resistance | interventions — Ultrasonography; Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — biobank 10 ml EDTA for DNA extraction
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- NAFLD + type 1 diabetes: type 1 diabetes patient with NAFLD on screening
  Interventions: Diagnostic Test: ultrasound; Diagnostic Test: elastography; Diagnostic Test: controlled attenuation parameter (CAP); Diagnostic Test: FLI; Diagnostic Test: FIB-4; Diagnostic Test: NFS
- noNAFLD + type 1 diabetes: type 1 diabetes patient without NAFLD on screening
  Interventions: Diagnostic Test: ultrasound; Diagnostic Test: elastography; Diagnostic Test: controlled attenuation parameter (CAP); Diagnostic Test: FLI; Diagnostic Test: FIB-4; Diagnostic Test: NFS

INTERVENTIONS:
Diagnostic Test: ultrasound — ultrasound to check for NAFLD according to Saverymuttu criteria
Diagnostic Test: elastography — elastography to compare liver stiffness indices
Diagnostic Test: controlled attenuation parameter (CAP) — CAP is a non-invasive additive on Fibroscan (trademark) which can quantify hepatic steatosis
Diagnostic Test: FLI — the FLI is a score panel designed to screen for NAFLD
Diagnostic Test: FIB-4 — the FIB-4 is a score panel designed to screen for significant fibrosis
Diagnostic Test: NFS — the NFS is a score panel designed to screen for significant fibrosis

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is a condition characterized by intrahepatic fat accumulation. It is closely related to insulin resistance. To date, it remains unclear whether NAFLD is common in patients with type 1 diabetes or if NAFLD translates into an increased health burden in this population. Screening for NAFLD is challenging due to the limitations of non-invasive diagnostic tools.

Liver biopsy remains the gold standard but is not suited for routine screening or clinical studies. Therefore, there is a great demand for accurate non-invasive screening tools that can not only diagnose but also stage NAFLD. This study aims to generate a large cohort of thoroughly characterized type 1 diabetes patients screened for NAFLD using multiple non-invasive tools including MRI, ultrasound, controlled attenuation parameter, and score panels. We aim to generate a biobank to promote a research collaboration network in the field of non-invasive diagnosis of NAFLD.

A secondary endpoint is to investigate the potential correlation between the presence of NAFLD and the occurrence of micro-or macrovascular complications in patients with diabetes.

DETAILED DESCRIPTION:
This study aims to characterize and follow a thoroughly characterized cohort of adult type 1 diabetes patients free from secondary liver disease due to excessive alcohol usage, viral hepatitis, alfa-1 antitrypsin deficiency, Wilson's disease or steatogenic or hepatotoxic drug use.

The investigators will screen for NAFLD and fibrosis using multiple non-invasive techniques including

* ultrasound
* controlled attenuation parameter
* fatty liver index
* human steatosis index
* transient elastography
* FIB-4
* NAFLD fibrosis score
* NASH algorithm based on multiple parameters

Subjects will be screened for microvascular and microvascular complications with:

* ECG
* microfilament examination
* 24hour urine collection for microalbuminuria
* serum kidney test (creatinine, eGFR)
* fundoscopy
* peripheral arterial pulsation palpation

The investigators will subsequently thoroughly characterize various metabolic and anthropometric parameters and document any microvascular or macrovascular complications.

The patients will be annually rescreened for both NAFLD-related as cardiovascular variables. Therefore this study will assess the correlation between NAFLD, cardiovascular risk, and type 1 diabetes in a prospective manner.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Adult age
* Informed consent given

Exclusion Criteria:

* Secondary liver disease
* Excess alcohol usage
* Pregnancy
* Use of steatogenic medication
* Active cancer or oncological treatment
* History of organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult type 1 diabetes patients followed in the outpatient diabetes clinic of the Antwerp University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD in type 1 diabetes: percentage of patients with indices of liver steatosis and/or NASH and/or fibrosis. | one year
  Determination of the cross-sectional prevalence of NAFLD in a cohort of type 1 diabetes patient (population size approximately 1000 subjects) according to ultrasound criteria, FLI≥60, HSI≥36, controlled attenuation parameter >215dB/m (M-probe) or ≥250 dB/m (XL probe) and MRI-PDFF >5% hepatocyte steatosis (reference method). All measures will be performed in a combined and standardized protocol to explore their diagnostic accuracy (see outcome 4).
Incidence of NAFLD in type 1 diabetes. | five years
  Incidence of NAFLD in type 1 diabetes determined by new cases of NAFLD according to ultrasound criteria, FLI≥60, HSI≥36, controlled attenuation parameter >215dB/m (M-probe) or ≥250 dB/m (XL probe) or MRI-PDFF >5% hepatocyte fat infiltration (reference method)
correlation of NAFLD with microvascular and macrovascular complications in type 1 diabetes mellitus: odds ratio to have prevalent complications in NAFLD and diabetes compared to diabetes without NAFLD | one year
  The correlation between indices of microvascular (neuropathy assessed by microfilament test, nephropathy assessed by microalbuminuria rate and retinopathy assessed by fundoscopic criteria) or macrovascular (non-fatal ischemic coronary disease, non-fatal cerebrovascular disease, non-fatal peripheral artery disease, or mortality due to cardiovascular disease) complications will be compared between groups with and without NAFLD as determined by the abovementioned screening tools.
Association of NAFLD with microvascular and macrovascular complications in type 1 diabetes mellitus: odds ratio to develop in NAFLD and diabetes compared to diabetes without NAFLD in subjects with no prior complications | five years
  The association between indices of microvascular (neuropathy assessed by microfilament test, nephropathy assessed by microalbuminuria rate and retinopathy assessed by fundoscopic criteria) or macrovascular (non-fatal ischemic coronary disease, non-fatal cerebrovascular disease, non-fatal peripheral artery disease or mortality due to cardiovascular disease) complications will be assessed between groups with and without NAFLD, but all without prior micro- or macrovascular disease as determined by the abovementioned screening tools.

SECONDARY OUTCOMES:
Diagnostic accuracy of non-invasive tools for NAFLD in type 1 diabetes: comparison of AUROC and diagnostic accuracy | five years
  The investigators will compare the abovementioned non-invasive tools to diagnose and grade liver steatosis and fibrosis with the predefined gold standard (MRI-PDFF for steatosis and magnetic resonance elastography for fibrosis). Correlations and agreement statistics will be performed for each index. Using regression analysis, a new specific algorithm will be developed based on cohort-specific cutoffs. Using longitudinal data, a prediction score will be determined to predict NAFLD occurrence or NAFLD progression.
Natural history of NAFLD in type 1 diabetes | five years
  Timewise description of the progression of quantitative indices of liver steatosis and fibrosis on the abovementioned tools (ultrasound, score systems, elastography) to assess the natural evolution of NAFLD. Every year this assay will be performed. MRI-PDFF will be performed in 5 years as a reference method to mark the five-year follow-up window

CONTACTS AND LOCATIONS:
Overall Officials: Christophe De Block, M.D., PhD, Principal Investigator — Universiteit Antwerpen; Sven Francque, M.D., PhD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
monocentric study

REFERENCES:
- [Background] de Vries M, Westerink J, Kaasjager KHAH, de Valk HW. Prevalence of Nonalcoholic Fatty Liver Disease (NAFLD) in Patients With Type 1 Diabetes Mellitus: A Systematic Review and Meta-Analysis. J Clin Endocrinol Metab. 2020 Dec 1;105(12):3842-53. doi: 10.1210/clinem/dgaa575. PMID 32827432
- [Background] Tana C, Ballestri S, Ricci F, Di Vincenzo A, Ticinesi A, Gallina S, Giamberardino MA, Cipollone F, Sutton R, Vettor R, Fedorowski A, Meschi T. Cardiovascular Risk in Non-Alcoholic Fatty Liver Disease: Mechanisms and Therapeutic Implications. Int J Environ Res Public Health. 2019 Aug 26;16(17):3104. doi: 10.3390/ijerph16173104. PMID 31455011
- [Background] European Association for the Study of the Liver (EASL); European Association for the Study of Diabetes (EASD); European Association for the Study of Obesity (EASO). EASL-EASD-EASO Clinical Practice Guidelines for the management of non-alcoholic fatty liver disease. J Hepatol. 2016 Jun;64(6):1388-402. doi: 10.1016/j.jhep.2015.11.004. Epub 2016 Apr 7. No abstract available. PMID 27062661
- [Background] Ismaiel A, Dumitrascu DL. Cardiovascular Risk in Fatty Liver Disease: The Liver-Heart Axis-Literature Review. Front Med (Lausanne). 2019 Sep 13;6:202. doi: 10.3389/fmed.2019.00202. eCollection 2019. PMID 31616668
- [Background] De Block CEM, Shivalkar B, Goovaerts W, Brits T, Carpentier K, Verrijken A, Van Hoof V, Parizel PM, Vrints C, Van Gaal LF. Coronary artery calcifications and diastolic dysfunction versus visceral fat area in type 1 diabetes: VISCERA study. J Diabetes Complications. 2018 Mar;32(3):271-278. doi: 10.1016/j.jdiacomp.2017.11.008. Epub 2017 Nov 28. PMID 29310998
- [Background] Hampson SJ. Nursing interventions for the first three postpartum months. J Obstet Gynecol Neonatal Nurs. 1989 Mar-Apr;18(2):116-22. doi: 10.1111/j.1552-6909.1989.tb00474.x. PMID 2709179